CLINICAL TRIAL: NCT04382248
Title: Next Generation Self Management: The Integration of a Mobile App Platform With Biomarkers in Kidney Transplantation
Brief Title: The Integration of a Mobile App Platform With Biomarkers in Kidney Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: CareDx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pro00104469
Record Dates: First submitted 2020-05-05; First posted 2020-05-11 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Medication Compliance
Keywords: kidney transplant; teens; mobile app
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Group (Experimental): An app for tracking medications, receiving personal coaching and educational material
  Interventions: Other: Smartphone App; Behavioral: Tailored education
- Control Group (Active Comparator): An app for tracking medications
  Interventions: Other: Smartphone App

INTERVENTIONS:
Other: Smartphone App — An app for monitoring medications, blood pressure, exercise, healthy eating
Behavioral: Tailored education — in-person coaching
  Arms: Interventional Group

SUMMARY:
The purpose of this study is to examine the feasibility and acceptability of a mobile app to improve self-management skills and medication adherence in kidney transplantation, to assess the clinical benefit of mobile app in combination with tailored coaching using text messaging to enhance patient activation, self-management and medication adherence and to determine whether immunological biomarkers such as cell-free DNA and donor specific antibodies are associated with self-management and medication adherence.

ELIGIBILITY:
Inclusion Criteria:

* 1) age 12-40 kidney transplant recipients with stable kidney function at least one month from the time of transplantation
* 2) have and use a smartphone
* 3) patients without pre-formed antibodies

Exclusion Criteria:

* 1) Patients <12 or >40
* 2) patient with pre-existing antibodies
* 3) patients with rejection at the time of enrollment
* 4) patients without a smartphone
* 5) patients with developmental delay or psychological impairment and unable to use an app

Ages: 12 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Change in patient activation scores as measured by Patient Activation Measure | baseline, 3 months, 6 months
  0-100 scale that segments patients into one of four activation levels
Change in self-management as measured by Partners In Health survey | baseline, 3 months, 6 months

SECONDARY OUTCOMES:
Medication adherence as measured by self-tracking | up to 6 months
Medication adherence as measured by blood levels | up to 6 months
Presence of cell-free DNA | up to 6 months
Presence of donor-specific antibodies | up to 6 months
Allograft function as measured by urine protein/creatinine ratio | up to 6 months
Allograft function as measured by serum creatinine | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Eileen Chambers, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No